CLINICAL TRIAL: NCT02403635
Title: A Single-centre, Open-label Study in Healthy Men to Investigate the Effect of Repeated Oral Doses of ASP2151 on the Pharmacokinetics of Midazolam in Healthy Men
Brief Title: Drug-Drug Interaction Study: ASP2151 and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho Europe Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M522101-EU24
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: HSV; Herpes; volunteers; drug-drug interaction
MeSH Terms: conditions — Herpes Simplex | interventions — Midazolam; ASP2151

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Midazolam + ASP2151 (Other): 400 mg ASP2151 followed by 7.5 mg midazolam
  Interventions: Drug: Midazolam; Drug: ASP2151

INTERVENTIONS:
Drug: Midazolam
  Other Names: Midazolam-ratiopharm
Drug: ASP2151

SUMMARY:
CYP3A4 is involved in the metabolism of many drugs. So, it is important to assess in vivo the induction effect of ASP2151 on that enzyme to determine the extent of any possible drug interactions. The aim of this trial is to investigate the potential for interaction of ASP2151 with the CYP3A4 probe substrate midazolam.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (Quetelet index) in the range 18.0-30.9.
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
* Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
* Willingness to give written consent to have data entered into The Overvolunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
* Any of the following liver function tests higher than 1.5 times the ULN at the screening visit: aspartate aminotransferase (AST), alanine aminotransferase (ALT), ALP, bilirubin, gamma glutamyl transpeptidase (gamma-GT).
* Platelet counts outside normal limits (129,000-346,000/µL).
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
* Clinically significant impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
* Presence or history of sleep apnoea or myasthenia gravis.
* History of bleeding diathesis.
* Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines.
* Presence or history of severe adverse reaction to any drug, history of multiple drug allergies (multiple defined as >3), or sensitivity to trial medication.
* Use, during the 28 days before the first dose of trial medication, of any prescription medicine, or any other medicine or herbal remedy (such as St John's wort) known to interfere with the CYP3A4, CYP2C19, CYP2C8 or CYP2C9 metabolic pathways.
* Use, during the 7 days before the first dose of trial medication, of any over the counter medicine, with the exception of paracetamol (acetaminophen).
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or intake of more than 21 units of alcohol weekly or more than 5 cigarettes daily.
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40_100 beats/min. However, if the investigator deems the result to be not clinically significant the subject may be included.
* Possibility that the volunteer will not cooperate with the requirements of the protocol.
* Evidence of drug abuse on urine testing.
* Positive test for hepatitis B, hepatitis C, HIV1 or HIV2.
* Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
* Objection by General Practitioner (GP) to volunteer entering trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Dr Kempeni, Study Director — Maruho Europe Ltd
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in United Kingdom from 18-March 2015 to 28-May 2015
Groups:
- Midazolam + ASP2151: 400 mg ASP2151 followed by 7.5 mg midazolam
  Midazolam
  ASP2151
Period: Overall Study
Arm/Group | Midazolam + ASP2151
Started | 27
Screening (28 Days) | 27
Received the First Dose | 18
Completed | 18
Not Completed | 9
Not completed — Not eligible | 9

BASELINE CHARACTERISTICS:
Arm/Group | Midazolam + ASP2151
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: year] | 30.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of Midazolam
Time Frame: prior to initial dose of Day 1 and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 h after dosing on Day 1, Days 12, 19 and 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Day 1; Day 19; Day 26: 7.5 mg midazolam alone
- Day 12: 7.5 mg midazolam with 400 mg ASP2151
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng/mL | 34.5 (21.2) | 23.4 (32.5) | 38.8 (23.1) | 36.8 (41.4)

2. Primary Outcome: Time of Peak Concentration (Tmax) of Midazolam
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
h | 0.5 [0.50 to 1.52] | 0.5 [0.25 to 150] | 0.5 [0.50 to 1.50] | 0.5 [0.28 to 2.00]

3. Primary Outcome: Area Under Concentration-Time Curve Extrapolated to Infinite Time (AUC0-∞) of Midazolam
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
h*ng/mL | 113.1 (28.1) | 58 (29.2) | 124.4 (31.7) | 122.1 (37.3)

4. Primary Outcome: Half-life (t1/2) of Midazolam
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
h | 4.2 (37) | 3.3 (52.7) | 4.3 (43.7) | 4.1 (52.3)

5. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Refer to the result of adverse event.
Time Frame: Up to 32 days after the last dose
Measure: Number; unit: participants
Groups:
- All Subjects: All subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 18
participants
  Non-serious adverse event | 18
  serious adverse event | 0

6. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of 1-hydroxymidazolam
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
ng/mL | 15.7 (33.2) | 15.9 (40.9) | 14.9 (35) | 14.2 (59.3)

7. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of 1-hydroxymidazolam
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
h | 0.5 [0.50 to 1.52] | 0.5 [0.25 to 150] | 0.5 [0.50 to 1.50] | 0.5 [0.28 to 1.50]

8. Other Pre Specified Outcome: Area Under Concentration-Time Curve up to Last Non-zero Value (AUC0-tn) of 1-hydroxymidazolam
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
h*ng/mL | 44 (30.3) | 39 (32.3) | 42.2 (31.3) | 40.4 (36.5)

9. Other Pre Specified Outcome: Half-life (t1/2) of 1-hydroxymidazolam
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
h | 3.8 (39.7) | 3.1 (47.4) | 3.5 (35.4) | 3.3 (42)

10. Other Pre Specified Outcome: Trough Plasma Concentration (Ctrough) of ASP2151
Time Frame: Days 5 to 12
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Day 5: Day 5 pre-dose
- Day 6: Day 6 pre-dose
- Day 7: Day 7 pre-dose
- Day 8: Day 8 pre-dose
- Day 9: Day 9 pre-dose
- Day 10: Day 10 pre-dose
- Day 11: Day 11 pre-dose
- Day 12: Day 12 pre-dose
Arm/Group | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | Day 10 | Day 11 | Day 12
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 18
ng/mL | 277.6 (73.47) | 265.7 (64.57) | 238.9 (65.6) | 240.7 (67.73) | 223.9 (63.68) | 228.5 (67.44) | 209.7 (66.47) | 214.2 (50.89)

11. Other Pre Specified Outcome: Peak Plasma Concentration (Cmax) of ASP2151
Time Frame: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 h after dosing on Day 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Day 12
Number analyzed (Participants) | 18
ng/mL | 1761.4 (37.9)

12. Other Pre Specified Outcome: Time of Peak Concentration (Tmax) of ASP2151
Time Frame: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 h after dosing on Day 12
Measure: Median (Full Range); unit: h
Arm/Group | Day 12
Number analyzed (Participants) | 18
h | 3 [1.00 to 5.00]

13. Other Pre Specified Outcome: Area Under Concentration-Time Curve Over the Dosing Interval (AUC0-tau) of ASP2151
Time Frame: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 h after dosing on Day 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 12
Number analyzed (Participants) | 18
h*ng/mL | 17167 (31.7)

14. Other Pre Specified Outcome: Area Under Concentration-Time Curve Extrapolated to Infinite Time (AUC0-∞) of ASP2151
Time Frame: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 h after dosing on Day 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 12
Number analyzed (Participants) | 18
h*ng/mL | 19334.2 (31.7)

15. Other Pre Specified Outcome: Half-life (t1/2) of ASP2151
Time Frame: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 h after dosing on Day 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Day 12
Number analyzed (Participants) | 18
h | 7.3 (12)

16. Other Pre Specified Outcome: Apparent Volume of Distribution (Vd/F) of ASP2151
Time Frame: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 h after dosing on Day 12
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Day 12
Number analyzed (Participants) | 18
L | 225.9 (65.66)

17. Other Pre Specified Outcome: Apparent Total Body Clearance (CL/F) of ASP2151
Time Frame: pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 h after dosing on Day 12
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Day 12
Number analyzed (Participants) | 24
L/h | 21.61 (6.35)

18. Other Pre Specified Outcome: Area Under Concentration-Time Curve up to Last Non-zero Value (AUC0-tn) of Midazolam
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
h*ng/mL | 111 (28) | 56.7 (28.8) | 121.9 (30.7) | 118.9 (36.2)

19. Other Pre Specified Outcome: Apparent Volume of Distribution (Vd/F) of Midazolam
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
L | 406.5 (46.3) | 622 (47) | 370.8 (43.1) | 366.6 (41)

20. Other Pre Specified Outcome: Apparent Total Body Clearance (CL/F) of Midazolam
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Day 1 | Day 12 | Day 19 | Day 26
Number analyzed (Participants) | 18 | 18 | 18 | 18
L/h | 444 (187.33) | 679.1 (276.5) | 401.3 (163.74) | 394 (153.76)

ADVERSE EVENTS:
Time Frame: Up to 32 days after the last dose
Groups:
- Midazolam: 7.5 mg midazolam
- ASP2151 After Midazolam: 400 mg ASP2151 after 7.5 mg midazolam
- Midazolam With ASP2151: 7.5 mg midazolam with 400 mg ASP2151
Arm/Group | Midazolam | ASP2151 After Midazolam | Midazolam With ASP2151 | Total
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 17/18 | 4/18 | 17/18 | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam (N=18) | ASP2151 After Midazolam (N=18) | Midazolam With ASP2151 (N=18) | Total (N=18)
Somnolence (Nervous system disorders) | 17 | 0 | 17 | 18
Headache (Nervous system disorders) | 0 | 1 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Catheter site inflammation (General disorders) | 1 | 0 | 0 | 1
Energy increased (General disorders) | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Lip haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No